CLINICAL TRIAL: NCT02045420
Title: Vascular Abnormalities in Idiopathic Parkinson's Disease
Acronym: IPD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Saskatchewan (Other)
Responsible Party: Sponsor
Other Study IDs: BIO13-204
Record Dates: First submitted 2013-12-11; First posted 2014-01-24 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Idiopathic Parkinson's Disease
Keywords: Idiopathic Parkinson's Disease; Magnetic Resonance Imaging; MR Venography; Flow Quantification; Susceptibility Weighted Imaging
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal Participants: The investigators will use "normal" age-matched volunteers to compare against the Idiopathic Parkinson's Disease Patients
- Idiopathic Parkinson's Disease Patients: The investigators will observe the MR scans to determine the vascular flow, brain lesions and brain iron levels in this group.

SUMMARY:
The purpose of this study is to use non-invasive Magnetic Resonance Imaging (MRI) scans to investigate venous insufficiency, brain iron levels and white matter hyperintensities (WMHs) to determine if there is direct correlation with Idiopathic Parkinson's Disease (IPD).

Idiopathic Parkinson's disease (IPD) is the second most common neurodegenerative disease after Alzheimer's disease and it affects roughly 0.1% to 0.3% of the population. The risk of having IPD increases with age and the median onset age is about 60 years. The etiology of IPD remains unknown. Generally, Parkinson's patients show a reduction of dopamine levels in the deep grey matter of the brain over time. Many clinically diagnosed cases of IPD are associated with white matter hyperintensities (WMH) and elevated brain iron levels. Furthermore, in the last few years there has been an increasing interest in the role of veins in neurodegenerative diseases. More attention has been paid to the extracranial veins as being potential sources of venous hypertension. The obstructed veins are thought to cause venous insufficiency. By using MRI techniques, the investigators can not only obtain qualitative vascular information but also quantitative arterial and venous blood flow measurements.

DETAILED DESCRIPTION:
Experimental plans: All patients and controls will consent to be subjects in this study. Data will be collected on the Siemens Skyra 3T scanner at the University of Saskatchewan using a 16 channel head/neck coil arrangement. The investigators main approach in this research is to collect MR data on the vasculature in the brain and neck, the iron content in the brain, and standard anatomical scans for 20 patients with idiopathic Parkinson's disease and 10 age matched normal subjects. MR venography, flow quantification and susceptibility weighted imaging will be used.

Anatomic MR venography (MRV): Contrast enhanced MRV is widely regarded as the optimal method for evaluation of disease involving the dural venous sinuses. It is an accurate, reliable and robust method for assessing sino-venous pathology such as thrombosis and tumor invasion. MRV is also able to demonstrate pathology involving larger cerebral veins. The investigators will be able to record both anatomic variants as well as any stenosis. Extracranially, the investigators will look for any significant variants or stenosis affecting the jugular venous system, the vertebral venous system and the azygous system. Data will be analyzed to separately display and evaluate the structure of arteries and veins in the head and neck. The maximum intensity projection (MIP) of the whole series will be generated in the coronal view. The major arteries will be evaluated as well as major veins of interest for the structural analysis including the transverse sinuses, the internal and external jugular veins, vertebral veins and deep cervical veins which usually serve as collaterals in case of flow abnormalities in the jugular veins. Cross sectional areas (CSA) of suspicious stenotic regions will also be measured to validate whether the variation seen in these CSA are veins stenosis or not.

Flow quantification (FQ): Pathological change in cerebrospinal venous drainage will be reflected by upstream disturbance of venous flow. Phase contrast MR flow techniques allow the investigators to interrogate venous flow. By applying FQ techniques to the dural venous sinuses, investigators hope to characterize the interplay between anatomic venous obstruction and pathologically altered drainage. By understanding this relationship, the investigators can gain deeper insight into the mechanism by which cerebrospinal venous insufficiency interacts with iron homeostasis mechanisms and ultimately with the pathogenesis of Parkinson's disease. Dural sinus hemodynamics can be studied non-invasively with phase contrast FQ. The phase contrast flow quantification (PCFQ) images will be used to analyze the through-plane cerebral spinal fluid in the neck (C2/C3 level), as well as blood flow in the neck (C2/C3 and C6/C7 levels), the superior sagittal sinus (SSS), both left and right transverse sinus, the straight sinus, both the extra cranial jugular and vertebral veins and Dural Sinus. Areas of interest will be drawn around the veins and arteries of interest and flow will be calculated over a full cardiac cycle. Thirty time points will be collected for each cardiac cycle by using a retroactive pulse trigger. The vessels of interest will include: the internal and external jugular veins (IJVs, EJVs), vertebral veins, deep cervical veins, common carotid arteries and vertebral arteries. The investigators will be evaluating the integrated flow, the average velocity, the volume flow rate, as well as negative and positive flow rate. This will be assessed in the cervical arteries to compare the inflow and outflow of the brain. Abnormalities may be identified by stressing the system, i.e., with a breath hold. Finally a large number of quantitative measures will be made on all the arteries and veins in the neck to assess both individual variants and total flow in the brain.

Measuring Iron in the basal ganglia and thalamus using Susceptibility Weighted Imaging (SWI): A presence of iron not only in lesions, but now more importantly in the basal ganglia and thalamus has been shown in IPD patients. The latter shows iron build up at the confluence of the draining veins in these areas. SWI can be run to show iron deposition in several areas of interest within the brain. SWI has very high spatial resolution and is an optimal method to study the small internal cerebral venous system. The ability to measure the amount of non-heme iron in the brain will facilitate a better understanding of the disease progression and may help in predicting the treatment outcome. Iron deposition will be evaluated from the SWI images. To measure iron content in grey matter, investigators will look at iron in the following eight regions: caudate nucleus, globus pallidus, putamen, thalamus, pulvinar thalamus (as it appears to be affected much before the rest of the thalamus), substantia nigra, red nucleus and dentate nucleus. For each deep gray matter structure, two major regions of interest will be analyzed: the entire object drawn manually and the region-of-interest that has much higher iron content. The investigators will provide the following information for these regions: iron content in the abnormal part of the structure (the investigators refer to this as the high iron content region); the area of this region; the average iron per pixel in this region; and also the investigators will quote the same three values for the total iron in these structures.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's Disease

Exclusion Criteria:

* Not MRI Compatible
* Diabetes
* Hypertension or Cardiac disease
* History of a Stroke
* Cardiac Pacemaker
* Have had Surgery for an Aneurysm
* Major Surgery within the last 8 weeks
* Claustrophobia
* Pregnant or Nursing

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be comprised of patients with Idiopathic Parkinson's Disease and Age-Matched Normal Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2013-12; Primary Completion 2016-10 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Measurement of Vascular Flow within the Internal Jugular Veins(IJVs), External Jugular Veins(EJVs) and Dural Sinus | MRI Baseline Scan: Not a Longitudinal Study
  Vascular Flow Rates within the head and neck will be measured using the MRI Flow Quantification tool. There is specific interest to correlate flow in the Dural Sinus, IJVs and EJVs and compare the measured flows with each participant's Unified Parkinson's Disease Rating Scale (UPDRS) Score.

SECONDARY OUTCOMES:
Measurement of Brian Iron using MRI Susceptibility Weighted Imaging Iron Quantification tools | MRI Baseline Scan: Not a Longitudinal Study
  Brain Iron levels within the Red Nuclei, Substantia Nigra, Globus Pallidus, Putamen, Caudate Nucleus and Thalamus will be measured. Given that Brain Iron levels increase with age, there is specific interest to correlate age dependent Brain Iron Levels to each participant's Unified Parkinson's Disease Rating Scale (UPDRS) Score.

OTHER OUTCOMES:
Quantity and size measurement of White Matter Hyperintensities (WMHs) | MRI Baseline Scan: Not a Longitudinal Study
  The number and size of White Matter Hyperintensities will be measured using the MRI -MPRAGE data. There is specific interest in determining if there is a correlation between WMHs and each participant's Unified Parkinson's Disease Rating Scale (UPDRS) Score.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Szkup, MD, Principal Investigator — University of Saskatchewan; Paul Babyn, MD, Study Director — University of Saskatchewan
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada